CLINICAL TRIAL: NCT06660017
Title: Ketamine Oral Rinse in the Management of Oral Mucositis in Head and Neck Cancer Patients Undergoing Radiation Therapy
Brief Title: Head and Neck Cancer Patients With Oral Mucositis Treated With Ketamine Oral Rinse
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OU-SCC-KORAL
Record Dates: First submitted 2024-10-24; First posted 2024-10-26 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Head and Neck Cancer
Keywords: Head and Neck Cancer; Ketamine; Oral Rinse; Radiation
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Ketamine

STUDY DESIGN:
Intervention Model Description: There will be a control group and an intervention group in this study. The control group will receive an unmedicated syrup solution in addition to standard treatment for oral mucositis. The intervention group will receive ketamine oral rinse in addition to standard treatment for oral mucositis.
Who Masked: Participant
Masking Description: The principal investigator and pharmacist will be the only ones who are aware of whom gets which arm of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Control Group (Placebo Comparator): Topical unmedicated syrup base + any standard treatment for oral mucositis.
  Interventions: Drug: Placebo
- Intervention Group (Experimental): Topical ketamine in syrup + any standard treatment for oral mucositis.
  Interventions: Drug: Ketamine Topical

INTERVENTIONS:
Drug: Placebo — Patients in this arm will receive unmedicated syrup solution dispensed as 20mg/5ml 4 times a day in addition to receiving one of the following standard treatments; Magic Mouthwash, saliva substitute rinses, over-the-counter remedies including honey or salt and soda rinses, non-steroidal anti-inflammatory drugs (NSAIDS), or opioid medications.
  Arms: Control Group
Drug: Ketamine Topical — Patients in this arm will receive ketamine oral rinse dispensed as 20mg/5ml 4 times a day in addition to receiving one of the following standard treatments; Magic Mouthwash, saliva substitute rinses, over-the-counter remedies including honey or salt and soda rinses, non-steroidal anti-inflammatory drugs (NSAIDS), or opioid medications.
  Arms: Intervention Group

SUMMARY:
This 2-arm phase II study proposes to determine the efficacy of ketamine oral rinse in pain relief from mucositis in head and neck cancer patients undergoing radiation treatment.

DETAILED DESCRIPTION:
Patients with histologically proven head and neck cancer undergoing radiation or concurrent chemoradiation as part of their treatment plan, will either receive ketamine oral rinse or unmedicated oral rinse to use 4 times a day if they develop oral mucositis during their radiation.

Patients will be monitored during treatment and up to 30 days after and will utilize a pain diary to document daily.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent signed and dated by the patient prior to the performance of the study-specific procedure.
2. At least 18 years-of-age at the time of signature of the informed consent form (ICF).
3. Patients with histologically proven HNSCC undergoing radiation of concurrent chemoradiation as part of their treatment plan.
4. Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0, 1, or 2.
5. The patients has received at least one radiation treatment for (HNSCC) the current disease.
6. CTCAE v. 5.0 grade 2 or greater oral cavity or pharyngeal mucositis documented to have developed after initiation of radiotherapy.
7. Males or female patients. Male patients with female partners of childbearing potential and female patients of childbearing potential are required to use two forms of acceptable contraception, including one barrier method, during their participation in the study and for 30 days following last dose. Male patients must also refrain from donating sperm during participation in the study.

Exclusion Criteria:

1. Inability to sign an informed consent form.
2. Any other malignancy diagnosed or treated within 10 years prior to enrollment.
3. Any documented hypersensitivity to ketamine.
4. Contraindication for ketamine use, including allergy.
5. Patients with schizophrenia, acute psychosis, or any psychiatric disorder that could be dangerous if exacerbated.
6. Women who are pregnant, nursing, or who plan to become pregnant while in the study and for at least <<6>> months after the last administration of study treatment.
7. Men who plan to father a child while in the study and for at least 6 months after the last administration of study treatment.
8. As judged by the Investigator, any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension, uncontrolled diabetes mellitus, active bleeding diatheses, or active infection including hepatitis B, hepatitis C, and human immunodeficiency virus. Screening for chronic conditions is not required.
9. Patients with a prior or concurrent malignancy whole natural history or treatment does not have potential to interfere with the safety or efficacy assessment of the investigational regimen should be included.
10. Psychological, familial, sociological, or geographical conditions that do not permit compliance with the protocol and/or follow-up procedures outlined in the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Number of patients who have altered pain response from mucositis in head and neck cancer undergoing radiation treatment from using ketamine oral rinse. | 6 months
  Review weekly questionnaires of patients who received ketamine oral rinse to assess if it helped with the pain of mucositis caused by the radiation in head and neck cancer patients.

SECONDARY OUTCOMES:
Number of patients whose dysphagia was decreased by the use of ketamine oral rinse among head and neck cancer patients undergoing radiation therapy. | 6 months.
  Dysphagia as assessed by MDADI.
Number of patients whose quality-of-life increased after the use of ketamine oral rinse among head and neck cancer patients undergoing radiation therapy. | 6 months
  Quality of life as assessed by FACT-HN.
Number of patients who need morphine prescription equivalent reductions as a result of using ketamine oral rinse. | 6 months
  Pain medication requirement measured in morphine equivalents.

CONTACTS AND LOCATIONS:
Overall Officials: Rusha Patel, MD, Principal Investigator — OU Health Stephenson Cancer Center
Locations (1):
- OU Health Stephenson Cancer Center, Oklahoma City, Oklahoma, United States